CLINICAL TRIAL: NCT05800808
Title: Exercise Induced Plasma Volume Expansion Lowers Cardiovascular Strain and Improves Cycling Time-trial Performance in Acute Normobaric Hypoxia
Brief Title: Exercise Induced Plasma Volume Expansion Lowers Cardiovascular Strain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Baptist University (Other)
Collaborators: High Point University (Other); United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Plasma Volume and Hypoxia
Record Dates: First submitted 2023-02-28; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Cardiac Output; Stroke Volume
Keywords: Hypervolemia; high intensity exercise; altitude exposure
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Exercise (Experimental): Vigorous cycling
  Interventions: Procedure: High Intensity Intervals
- Continuous Moderate Exercise (Active Comparator): Leisurely cycling
  Interventions: Procedure: Moderate Exercise

INTERVENTIONS:
Procedure: High Intensity Intervals — 8x4 min cycling bouts at 85% of VO2peak
  Arms: High Intensity Exercise
Procedure: Moderate Exercise — 81 minutes of cycling at 50% VO2peak
  Arms: Continuous Moderate Exercise

SUMMARY:
The goal of this observational study was to better understand the impact of increased plasma volume on later exercise in hypoxia. Investigators examined young, healthy, males who regularly participated in aerobic exercise.

Investigators first measured participant's response to exercise in hypoxia (simulated ~7,500 feet above sea level). The investigators then had participants either 1) undergo 1 bout of high intensity interval exercise or 2) undergo 1 bout of moderate, continuous exercise.

48 hours after the exercise, participants were again examined in hypoxia.

DETAILED DESCRIPTION:
A crossover design was utilized to assess the effects of exercise-induced plasma volume expansion on cycling performance in hypoxia. All participants completed a high intensity (HI) bout and control (CON) intervention in a counterbalanced order. The HI bout consisted of 8x4min cycling bouts at 85% of VO2peak with 4 min rest between intervals. CON consisted of cycling at 50% VO2peak. Two 15 km, self-paced cycling time trials (TT) were performed before and after each training intervention. The first TT occurred 5 days before the training intervention (HI or CON) and the second TT occurred 48 hours post intervention. Interventions were separated by 14 days to ensure sufficient washout of any training effect as data have suggested retention of expanded plasma volume may last for 7-14 days. During washout, participants were instructed to continue their normal exercise routine.

The investigators hypothesized that a single HI session would increase plasma volume and attenuate cardiovascular strain during exercise in hypoxia, as evidenced by reductions in HR and elevations in SV and Q. Furthermore, the investigators hypothesized that these changes would contribute to a reduced time-to-completion in a 15 km, self-paced cycling TT.

ELIGIBILITY:
Inclusion Criteria:

* Males age 18-38
* Exercise at least 3 times/week for at least 30 minutes/day for the past 3 months.

Exclusion Criteria:

* Frequent hot bath or sauna users
* Resided at altitude greater than 2,500 meters for >14 days.
* Cardiovascular or metabolic disease

Ages: 18 Years to 38 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Hemoglobin Concentration | through study completion, an average of 4 weeks
  measured through spectroscopy
Hematocrit Concentration | through study completion, an average of 4 weeks
  measured through hematocrit reader

SECONDARY OUTCOMES:
Time Trial Time | through study completion, an average of 4 weeks
  Time to complete 15 km
Cardiac Output | through study completion, an average of 4 weeks
  measured via impedance cardiography

CONTACTS AND LOCATIONS:
Locations (1):
- California Baptist University, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alexander JK, Hartley LH, Modelski M, Grover RF. Reduction of stroke volume during exercise in man following ascent to 3,100 m altitude. J Appl Physiol. 1967 Dec;23(6):849-58. doi: 10.1152/jappl.1967.23.6.849. No abstract available. PMID 6065055
- [Background] Beidleman BA, Staab JE, Muza SR, Sawka MN. Quantitative model of hematologic and plasma volume responses after ascent and acclimation to moderate to high altitudes. Am J Physiol Regul Integr Comp Physiol. 2017 Feb 1;312(2):R265-R272. doi: 10.1152/ajpregu.00225.2016. Epub 2016 Dec 30. PMID 28039191
- [Background] Berger NJ, Campbell IT, Wilkerson DP, Jones AM. Influence of acute plasma volume expansion on VO2 kinetics, VO2 peak, and performance during high-intensity cycle exercise. J Appl Physiol (1985). 2006 Sep;101(3):707-14. doi: 10.1152/japplphysiol.00154.2006. Epub 2006 May 11. PMID 16690793
- [Background] Brothers MD, Wilber RL, Byrnes WC. Physical fitness and hematological changes during acclimatization to moderate altitude: a retrospective study. High Alt Med Biol. 2007 Fall;8(3):213-24. doi: 10.1089/ham.2007.8308. PMID 17824822
- [Background] Chapman RF, Laymon AS, Levine BD. Timing of arrival and pre-acclimatization strategies for the endurance athlete competing at moderate to high altitudes. High Alt Med Biol. 2013 Dec;14(4):319-24. doi: 10.1089/ham.2013.1022. PMID 24377334
- [Background] Chapman RF, Stager JM, Tanner DA, Stray-Gundersen J, Levine BD. Impairment of 3000-m run time at altitude is influenced by arterial oxyhemoglobin saturation. Med Sci Sports Exerc. 2011 Sep;43(9):1649-56. doi: 10.1249/MSS.0b013e318211bf45. PMID 21311361
- [Background] Chapman RF, Stickford JL, Levine BD. Altitude training considerations for the winter sport athlete. Exp Physiol. 2010 Mar;95(3):411-21. doi: 10.1113/expphysiol.2009.050377. Epub 2009 Oct 16. PMID 19837773
- [Background] Coles MG, Luetkemeier MJ. Sodium-facilitated hypervolemia, endurance performance, and thermoregulation. Int J Sports Med. 2005 Apr;26(3):182-7. doi: 10.1055/s-2004-820989. PMID 15776333
- [Background] Coyle EF, Hopper MK, Coggan AR. Maximal oxygen uptake relative to plasma volume expansion. Int J Sports Med. 1990 Apr;11(2):116-9. doi: 10.1055/s-2007-1024774. PMID 1692570
- [Background] Fortney SM, Wenger CB, Bove JR, Nadel ER. Effect of blood volume on forearm venous and cardiac stroke volume during exercise. J Appl Physiol Respir Environ Exerc Physiol. 1983 Sep;55(3):884-90. doi: 10.1152/jappl.1983.55.3.884. PMID 6629925
- [Background] Fulco CS, Muza SR, Beidleman BA, Demes R, Staab JE, Jones JE, Cymerman A. Effect of repeated normobaric hypoxia exposures during sleep on acute mountain sickness, exercise performance, and sleep during exposure to terrestrial altitude. Am J Physiol Regul Integr Comp Physiol. 2011 Feb;300(2):R428-36. doi: 10.1152/ajpregu.00633.2010. Epub 2010 Dec 1. PMID 21123763
- [Background] Fulco CS, Rock PB, Cymerman A. Maximal and submaximal exercise performance at altitude. Aviat Space Environ Med. 1998 Aug;69(8):793-801. PMID 9715971
- [Background] Gillen CM, Lee R, Mack GW, Tomaselli CM, Nishiyasu T, Nadel ER. Plasma volume expansion in humans after a single intense exercise protocol. J Appl Physiol (1985). 1991 Nov;71(5):1914-20. doi: 10.1152/jappl.1991.71.5.1914. PMID 1761491
- [Background] Gillen CM, Nishiyasu T, Langhans G, Weseman C, Mack GW, Nadel ER. Cardiovascular and renal function during exercise-induced blood volume expansion in men. J Appl Physiol (1985). 1994 Jun;76(6):2602-10. doi: 10.1152/jappl.1994.76.6.2602. PMID 7928889
- [Background] Greenleaf JE, Looft-Wilson R, Wisherd JL, Jackson CG, Fung PP, Ertl AC, Barnes PR, Jensen CD, Whittam JH. Hypervolemia in men from fluid ingestion at rest and during exercise. Aviat Space Environ Med. 1998 Apr;69(4):374-86. PMID 9561285
- [Derived] Gorini Pereira F, Greenfield AM, Kuennen M, Gillum TL. Exercise induced plasma volume expansion lowers cardiovascular strain during 15-km cycling time-trial in acute normobaric hypoxia. PLoS One. 2024 Feb 2;19(2):e0297553. doi: 10.1371/journal.pone.0297553. eCollection 2024. PMID 38306343